CLINICAL TRIAL: NCT07184554
Title: Comparison of the Effectiveness of Lumbar Erector Spinae Plane Block and Lumbar Interlaminar Epidural Steroid Injection in Patients With Lumbar Disc Herniation.
Brief Title: Lumbar Disc Hernia, Erector Spinae Plane Block, Ilesi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Damla Yürük, Supervisor Investigator, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Ilesi block vs esp
Record Dates: First submitted 2025-09-10; First posted 2025-09-22 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Lumbar Disc Herniation
Keywords: espb, lesi, lumbar disc herniation
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- us-guided espb (Active Comparator): us-guided espb for ldh
  Interventions: Procedure: us-guided espb
- fl-guided Ilesi (Active Comparator): fl-guided Ilesi for ldh
  Interventions: Procedure: fl-guided Ilesi

INTERVENTIONS:
Procedure: us-guided espb — Hemodynamic monitoring is provided. The lumbar region where the procedure will be performed is cleaned with povidone iodine. Sterile draping is provided. For the lumbar erector spinae plane block application, a 5 Hz convex ultrasound probe is first placed sagittally over the desired level of the lumbar vertebra. After the spinous processes are visualized, the ultrasound probe is laterally shifted in the sagittal plane, first visualizing the laminae, then the facet joints, and finally the transverse processes. The erector spinae muscles are visualized over the transverse processes. The skin and subcutaneous tissue are then anesthetized with 2 cc of 2% lidocaine. A spinal needle is inserted from the anesthetized area in the same plane as the ultrasound probe (in plane) and contacts the relevant transverse process. Thanks to the real-time imaging advantage of ultrasound, a certain distance is maintained from the nerves and vascular structures. Once the appropriate location is reached, a m
  Arms: us-guided espb
Procedure: fl-guided Ilesi — For lumbar interlaminar epidural steroid injection, the anterior view of the desired level is obtained under fluoroscopy to visualize the relevant interlaminar epidural space. The skin and subcutaneous tissue are anesthetized with a local anesthetic. A paramedian approach is used to enter the target interlaminar space with an epidural needle using a negative pressure injector. The lateral view is checked using fluoroscopy. 2 cc of opaque material is administered, and its presence in the epidural space is confirmed from the lateral and anterior-posterior views. A mixture of steroid and local anesthetic (8 mg dexamethasone, 3 cc 5mg/ml bupivacaine, and SF for a total of 10 cc) is injected. The needle is removed in a controlled manner and the needle site is closed. After the procedure, patients are monitored in the recovery unit for 60 minutes and then transferred to the ward for follow-up. Patients who have completed their 1-hour follow-up in the ward are discharged.
  Arms: fl-guided Ilesi

SUMMARY:
The study is designed as an observational study. Patients who have been treated and completed treatment for lumbar discopathy in our clinic will be followed. Patients will not be divided into groups beforehand, and this will not cause changes to the treatment plan. Patients who have undergone fluoroscopy-guided lumbar interlaminar epidural steroid injection (LESI) and ultrasound-guided lumbar erector spinae plane block (LESP), routinely performed in our clinic for the treatment of back and leg pain due to lumbar disc herniation, will be compared to the effectiveness of these methods on pain at baseline before the procedure and at 2, 6, and 12 weeks afterward using the Visual Analogue Scale for Pain Relief (VAS) and Oswestry Disability Index (ODI). The baseline values will be recorded from the patient files and by request before the start of follow-up.

DETAILED DESCRIPTION:
Chronic low back pain (>3 months) is one of the chronic pain syndromes that most significantly impairs functionality. Lumbar disc herniation is one of the most common spinal degenerative conditions causing low back pain and radicular leg pain. Treatment options for this condition in pain clinics include minimally invasive treatments such as paravertebral plane blocks and epidural steroid injections. The use of interventional methods for low back pain has been increasing in recent years. The primary reason for this is the desire of patients who fail to achieve adequate relief with conservative treatment methods such as medical therapy and physical therapy to try relatively conservative methods before surgery. Two commonly used interventions for patients with lumbar disc herniation who do not respond to conservative treatment methods are fluoroscopy-guided LESI and ultrasound-guided LESP block, which we frequently perform in our clinic.

Patients who have undergone routine LESP and LESI in our clinic and who meet the inclusion criteria will be included in the study. Pain intensity and functionality will be assessed using the visual analog pain score and the Oswestry disability index.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic low back pain caused by L4-L5 and L5-S1 lumbar disc herniation accompanied by radicular pain, including those diagnosed by MRI, will be included.
* Patients with low back pain above VAS 5 for more than 6 weeks will be included.
* Failure of pain treatment with conservative methods such as analgesics and physical therapy

Exclusion Criteria:

* Patients who have previously undergone lumbar surgery,
* Patients with spinal deformity and stenosis,
* Patients with uncontrolled diabetes
* Patients allergic to the drugs to be used will not be included in the study.
* Presence of psychiatric comorbidity
* Local or systemic infection
* Coagulopathy
* Presence of rheumatological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-20 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) | Change from baseline to 2nd, 6th and 12th weeks after treatment
  VAS is a scale that can be used measuring pain. Scores range from 0 (no pain) to 10 (the worst pain)

SECONDARY OUTCOMES:
oswestry disability index | Change from baseline to 2nd, 6th and 12th weeks after treatment
  The Oswestry Disability Index is an index derived from the Oswestry Back Pain Questionnaire, which is used by clinicians and researchers to measure disability in terms of back pain and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Gevher Rabia Genc Perdecioğlu, Study Chair — Diskapi TRH
Locations (1):
- Etlik City Hospital, Ankara, Turkey (Türkiye)